CLINICAL TRIAL: NCT02769377
Title: Efficacy of Combination of Glucometer and Mobile-phone Based Data Transfer System on Glycemic Control in Patients With Diabetes
Brief Title: Glucometer and Mobile-phone Based Data Transfer System in Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, M.D., Ph.D., Taichung Veterans General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE15126B
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: diabetes, glucometer, mobile-phone
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): patients who decline or unable to do self-monitoring of blood glucose
- Breeze2 glucometer (Active Comparator): patients who do self-monitoring of blood glucose, but do not transfer data via mobile-phone
  Interventions: Device: Breeze2 glucometer
- Breeze2 glucometer and H2 (Experimental): patients who do self-monitoring of blood glucose and transfer data via mobile-phone
  Interventions: Device: Breeze2 glucometer; Device: Breeze2 glucometer and H2

INTERVENTIONS:
Device: Breeze2 glucometer — Breeze2 glucometer for self-monitoring of blood glucose
  Arms: Breeze2 glucometer; Breeze2 glucometer and H2
Device: Breeze2 glucometer and H2 — Breeze2 glucometer and Health2Sync Mobile App for data transfer
  Arms: Breeze2 glucometer and H2

SUMMARY:
To determine if glucometer combined with mobile-phone based data transfer system would be useful for patient diabetes to manage their glycemic control.

DETAILED DESCRIPTION:
Patients with diabetes who are advised by their providers to self-monitoring of blood glucose are eligible. Patients who decline or are not able to do self-monitoring of blood glucose will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with diabetes
2. Patients' providers advised self-monitor of blood glucose
3. Provided written informed consent.

Exclusion Criteria:

1. Patients had other medical condition that were considered not eligible by the medical team members

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | HbA1c change from baseline at month 3 and 6

SECONDARY OUTCOMES:
Hypoglycemia | event of hypoglycemia at month 3 and 6
  Hypoglycemia was defined as a glucose value less than 70 mg/dl, or with typical symptoms of hypoglycemia. The information of hypoglycemia will be collected at each site visit (every 1-2 month).

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Sheu, MD. Ph.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No